CLINICAL TRIAL: NCT01429597
Title: Fabry and Cardiomyopathy (FaCard) Epidemiological Study for the Analysis of Biomarkers and the Clinical Course of Patients With Fabry Disease and the N215S-mutation An Internationa,Multicenter, Epidemiological Study
Brief Title: Fabry and Cardiomyopathy (FaCard)
Acronym: FaCard
Status: Withdrawn | Type: Observational
Why Stopped: University of Rostock terminated participation in the study conduct; Study Sponsorship is moved to Centogene AG
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: FaCard06/2011
Record Dates: First submitted 2011-09-06; First posted 2011-09-07 (Estimated); Last update posted 2021-04-09 (Actual); Status verified 2020-04

CONDITIONS: Cerebrovascular Accident; Stroke, Acute; Cerebral Stroke
Keywords: Cerebrovascular Accident; Cerebrovascular Accident, Acute; Fabry Disease; Fabry´s Disease; Anderson-Fabry Disease; CVA (Cerebrovascular Accident); Stroke, Acute; Cerebral Stroke
MeSH Terms: conditions — Stroke; Fabry Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The laboratory examinations of the blood samples for measuring the lyso-Gb3-level will be done at the Laboratory of the Albrecht-Kossel-Institute, University of Rostock in collaboration with associated diagnostic laboratory partners. This laboratory offers an existing infrastructure, a highly standardized quality of the workflow, a short examination time of the samples and a long period of experiences in the assessment of the biological impact of mutations and polymorphism, as evidenced recently in the sifap1-study.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observation: All Patients with a diagnosis of Fabry disease with N215S

SUMMARY:
Primary objective and endpoint is the analysis of the long-term course of lyso-Gb3 and its clinical correlation to the progression of the cardiomyopathy in N215S-Fabry patients.

DETAILED DESCRIPTION:
Fabry disease is an X-linked lysosomal disorder that leads to excessive deposition of neutral glycosphingolipids in the vascular endothelium of several organs in the body. Progressive endothelial accumulation of glycosphingolipids accounts for the associated clinical abnormalities of skin, eye, kidney, heart, brain, and peripheral nervous system. Fabry disease manifesting predominantly in men. Female heterozygotes also present with features of Fabry disease. It is suggested that the mean age of hemizygotic men at the onset of symptomatic stroke is 29 - 34 years. The mean age of female heterozygotes at the onset of symptomatic strokes is 40 - 43 years.In Europe the prevalence of Fabry disease seems to be massively underrepresented; actual textbooks describe 1 per 40.000. However, recent data (Lin HY, et al., 2009) demonstrate the identification of eight different mutations in the alpha-galactosidase A (alpha-Gal A) gene in 110 027 newborns who were screened by assaying the alpha-Gal A activity followed by genetic analysis. Hwu and co-workers (2009) have shown in 90,288 male newborns screened for Fabry disease that 73 males had GLA gene mutations. Surprisingly, 86% had the c.936+919G>A (also called IVS4+919G>A) splice mutation. In contrast, screening 81,689 females detected two heterozygotes. Summarizing, newborn screening identified a surprisingly high frequency of Taiwanese males with Fabry disease (approximately 1 in 1,250), 86% having the IVS4+919G>A mutation previously found in later-onset cardiac phenotype patients.The late-onset mutation N215S is discussed to be a so-called cardiac variant (Perry Elliott, 2006; Eng et al., 1993, Sachdev et al., 2002). The prevalence of most mutations is low, i.e. Fabry disease spontaneously and individually inheriting so-called private mutations. However, there are some mutations that occur more frequent. Besides for instance R112H, A143T and R227X, also N215S belongs to this group (Dobrovolny et al., ASHG Abstract, 2008). The enzyme activity is only moderately affected, but hemizygous patients display a clearly decreased activity in leucocytes and fibroblasts.

In 2005, Young and colleagues (Acta Paediatr Suppl.) concluded that Gb3 is not an ideal biomarker using the example of N215S. All heterozygotes were unconspicuous and only 50% of the examined hemizygotes had increased levels. However, globotraosylceramid (lyso Gb3) seems to reveal all (genetically) found patients with a pathologically elevated level (with a mean of 1,17ng/ml (females) and 2,43ng/ml (males) respectively).

In a case study from 2004 (Meehan et al., American Journal of Kidney Diseases) was shown that a hemizygous male 75 years of age had a renal manifestation of mild proteinuria and a mildly decreased renal function due to high Gb3 accumulation in podocytes, to a lesser extent in tubular endothelial cells. Furthermore, he had mild congestive heart failure, a reduced left ventricular ejection fraction, and hypercholesterolemia. Thus, it is obvious that in Fabry patients with the N215S mutation disease progression can be mono- to oligosymptomatic, but show a tendency for the cardiac and renal phenotype rather than classical manifestation.

ELIGIBILITY:
Inclusion Criteria:

* All patients of both gender from 18 years of age with a diagnosis of Fabry disease with the mutation N215S
* Written informed consent from patient

Exclusion Criteria:

* Patients without a diagnosis of Fabry disease
* No written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Patients with a diagnosis of Fabry disease with N215S
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-07-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
analysis of the long-term course of lyso-Gb3 and its clinical correlation to the progression of the cardiomyopathy in N215S-Fabry patients | 24 month

CONTACTS AND LOCATIONS:
Overall Officials: Arndt Rolfs, Prof. Dr., Principal Investigator — CENTOGENE GmbH Rostock
Locations (1):
- University of Rostock, Albrecht-Kossel-Institute for Neuroregeneration, Rostock, Germany

IPD SHARING:
Plan to Share IPD: Undecided